CLINICAL TRIAL: NCT04087772
Title: Enhancing School-Based Violence Prevention Through Multilevel Racial/Ethnic Discrimination Intervention
Brief Title: Enhancing School-Based Violence Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00085255; 1R01MD013812-01 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Aggressive Childhood Behavior
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health-Enhanced PBIS (Active Comparator): Mental health-enhanced Positive Behavioral Interventions and Supports (PBIS-MH) integrates mental health into the three core elements of PBIS. 1) School-based mental health clinicians are included on leadership teams. 2) Data from teacher and student perceived school climate, as well as universal screening for aggression and mental health difficulties, are used to inform intervention decision-making. 3) Evidence-based mental health prevention and intervention practices are layered into PBIS' three-tiered continuum.
  Interventions: Behavioral: Mental Health Enhanced Positive Behavioral Interventions and Supports (PBIS-MH)
- Mental Health-Enhanced PBIS + RED (Experimental): PBIS-MH+RED involves the components of PBIS-MH integrated with racial/ethnic discrimination interventions (RED) to address multiple forms of school-based racial and ethnic discrimination. 1) Unintentional bias training for school personnel, involving teaching participants to conceptualize prejudice as well as strategies to reduce bias. 2) Unintentional bias training for students that is delivered in a classroom in a developmentally appropriate lesson format. 3) Vulnerable Decision Point process: Leadership teams are trained to reduce disparities in school discipline by a) using disaggregated student discipline data to identify particular settings or practices that are drivers for racial/ethnic disproportionality in a school and b) using iterative problem-solving to address these drivers. 4) Teacher stress reduction training where they are provided with strategies to reduce stress.
  Interventions: Behavioral: Mental Health Enhanced Positive Behavioral Interventions and Supports (PBIS-MH); Behavioral: Racial/Ethnic Discrimination Interventions (RED)

INTERVENTIONS:
Behavioral: Mental Health Enhanced Positive Behavioral Interventions and Supports (PBIS-MH) — Mental health-enhanced Positive Behavioral Interventions and Supports (PBIS-MH) integrates mental health into the three core elements of PBIS. 1) School-based mental health clinicians are included on leadership teams. 2) Data from teacher and student perceived school climate, as well as universal screening for aggression and mental health difficulties, are used to inform intervention decision-making. 3) Evidence-based mental health prevention and intervention practices are layered into PBIS' three-tiered continuum.
  Other Names: Interconnected Systems Framework
Behavioral: Racial/Ethnic Discrimination Interventions (RED) — Racial/Ethnic Discrimination Interventions are a set of components to address multiple forms of school-based racial and ethnic discrimination. 1) Unintentional bias training for school personnel, involving teaching participants to conceptualize prejudice as well as strategies to reduce bias. 2) Unintentional bias training for students that is delivered in a classroom in a developmentally appropriate lesson format. 3) Vulnerable Decision Point process: Leadership teams are trained to reduce disparities in school discipline by a) using disaggregated student discipline data to identify particular settings or practices that are drivers for racial/ethnic disproportionality in a school and b) using iterative problem-solving to address these drivers. 4) Teacher stress reduction training where they are provided with strategies to reduce stress.
  Arms: Mental Health-Enhanced PBIS + RED

SUMMARY:
The purpose of this study is to compare two versions of Mental Health Enhanced Positive Behavioral Interventions and Supports in reducing aggression in middle school students.

ELIGIBILITY:
Inclusion Criteria:

* for student participants: in 6th and 7th grades in a study school at study entry
* for teacher participants: teacher at a study school

Exclusion Criteria:

* .for student participants: intellectual disabilities, very limited reading abilities, or in foster care

Ages: 10 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4840 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in student report on aggression as measured by the Reactive and Proactive Aggression Survey | Fall of year 1 (average of October), spring of years 1 and 2 (average of May)
  The Reactive and Proactive Aggression Survey is a self-report instrument assessing how often the respondent has behaved aggressively towards other children over the past three months. Scores range from 0 (Never) to 5 (All of the time)
Mean change from baseline in teacher report on students' aggression as measured by the Teacher Report of Aggression | Fall of year 1 (average of October), spring of years 1 and 2 (average of May)
  The Teacher Report of Aggression is a teacher-report survey completed by teachers assessing a student's tendency to be aggressive. Scores range from 1 (Never) to 5 (All of the time)
Mean change from baseline in student aggression as measured by the number of Office Discipline Referrals per month | From first day of school in year 1 to last day of school in year 2
  Office Discipline Referrals are official school records recorded for each behavioral infraction warranting referral to the school office. Office Discipline Referrals for aggressive behavior (i.e. bullying, fighting, making threats) will be counted. The minimum score is 0 an there is no maximum score.

SECONDARY OUTCOMES:
Change from baseline in student report on discrimination from teachers as measured by the Adolescent Discrimination Index - Educational Discrimination Distress Subscale | Fall of year 1 (average of October), spring of years 1 and 2 (average of May)
  The Adolescent Discrimination Index is a self-report survey assessing the respondent's own experiences of racial/ethnic discrimination. The Education subscale assesses discrimination from school teachers.The respondent indicates whether they have experienced discrimination, either Yes or No. If the respondent selects Yes, they rate how upsetting the experience was with scores ranging from 1 (Not at all) to 5 (Extremely)
Change from baseline in student report on discrimination from peers as measured by the Adolescent Discrimination Index - Peer Discrimination Distress Subscale | Fall of year 1 (average of October), spring of years 1 and 2 (average of May)
  The Adolescent Discrimination Index is a self-report survey assessing the respondent's own experiences of racial/ethnic discrimination. The Peer subscale assesses discrimination from peers. The respondent indicates whether they have experienced discrimination, either Yes or No. If the respondent selects Yes, they rate how upsetting the experience was with scores ranging from 1 (Not at all) to 5 (Extremely)

CONTACTS AND LOCATIONS:
Locations (1):
- Name and state withheld to protect anonyminty of study site, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04087772/ICF_000.pdf